CLINICAL TRIAL: NCT04018885
Title: A Multi-center, Open, Randomized, Parallel Group Study to Assess Safety, Tolerance and Preliminary Efficacy of ALA for the Treatment of Moderate to Severe Acne Vulgaris
Brief Title: A Study on Safety and Preliminary Efficacy of ALA in Acne Vulgaris
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F0014-ALA-201809
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- ALA 2.5% 0.5h (Experimental): Topical application of 2.5% ALA for 0.5 hour
  Interventions: Drug: ALA 2.5%
- ALA 2.5% 1.5h (Experimental): Topical application of 2.5% ALA for 1.5 hours
  Interventions: Drug: ALA 2.5%
- ALA 2.5% 3h (Experimental): Topical application of 2.5% ALA for 3 hours
  Interventions: Drug: ALA 2.5%
- ALA 5% 0.5h (Experimental): Topical application of 5% ALA for 0.5 hour
  Interventions: Drug: ALA 5%
- ALA 5% 1.5h (Experimental): Topical application of 5% ALA for 1.5 hours
  Interventions: Drug: ALA 5%
- ALA 5% 3h (Experimental): Topical application of 5% ALA for 3 hours
  Interventions: Drug: ALA 5%
- ALA 10% 0.5h (Experimental): Topical application of 10% ALA for 0.5 hour
  Interventions: Drug: ALA 10%
- ALA 10% 1.5h (Experimental): Topical application of 10% ALA for 1.5 hours
  Interventions: Drug: ALA 10%
- ALA 10% 3h (Experimental): Topical application of 10% ALA for 3 hours
  Interventions: Drug: ALA 10%

INTERVENTIONS:
Drug: ALA 2.5% — Topical treatment for photodynamic therapy, after drug incubation subsequent illumination with red light (72 J/cm2). 4 treatments at an interval of 10 (± 4) days.
  Arms: ALA 2.5% 0.5h; ALA 2.5% 1.5h; ALA 2.5% 3h
Drug: ALA 5% — Topical treatment for photodynamic therapy, after drug incubation subsequent illumination with red light (72 J/cm2). 4 treatments at an interval of 10 (± 4) days.
  Arms: ALA 5% 0.5h; ALA 5% 1.5h; ALA 5% 3h
Drug: ALA 10% — Topical treatment for photodynamic therapy, after drug incubation subsequent illumination with red light (72 J/cm2). 4 treatments at an interval of 10 (± 4) days.
  Arms: ALA 10% 0.5h; ALA 10% 1.5h; ALA 10% 3h

SUMMARY:
The purpose of this study is to explore the safety, tolerability, and preliminary efficacy of ALA used with photodynamic therapy for the treatment of moderate to severe acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese male or female patients aged 18 - 40 years;
2. Grade III-IV facial acne vulgaris according to the Pillsbury International Improvement scale.;
3. All patients claimed to take effective contraception from 14 days before to 1 month after the end of the study, (among those who had used contraceptive two weeks prior to the study, the dosage of the drug should remain the same throughout the study) and had no fertility or donation of sperm/egg plan;
4. Informed consents were signed.

Exclusion Criteria:

1. Suffering with malignant tumors, cardiac, endocrine, blood, liver, immunity, metabolism, urinary system, lungs, nervous system, rheumatism / joint, psychology and kidney diseases;
2. Obviously abnormal liver and kidney function;
3. Suffering with allergy diseases; suspected or known to have porphyria; allergic to studying drugs and / or porphyrin; allergic to visible light; allergic constitution (allergic to two or more drugs, food or pollen);
4. Secondary acne patients, such as occupational acne or acne caused by corticosteroids;
5. Complicated with other obvious facial skin diseases such as actinic dermatitis, psoriasis, seborrheic dermatitis, eczema, skin tumors, etc;
6. Other diseases that may significantly affect the efficacy evaluation;
7. Pregnancy, lactation patients;
8. Exposed to systemic retinoids 2 months prior to the study (acitretin for 6 months);
9. Exposed to systemic antibiotics, glucocorticoids, spironolactone and other drugs for treating acne 4 weeks prior to the study; physical therapy for the treatment of acne;
10. Exposed to topical retinoids on the face 4 weeks prior to the study or topical antibiotics, glucocorticoids, and other topical treatment 2 weeks prior to the study;
11. Participated in other clinical trials 3 months prior to the study;
12. Other reasons that the investigator considered inappropriate for participation in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Success rate in Investigator's Global Assessment (IGA)(8wks) | 8 weeks after the last treatment
  Proportion of subjects with an assessment of clear or almost clear with at least a 2-grade improvement in IGA
Percent Changes From Baseline in Total Lesion Counts | 8 weeks after the last treatment
Number of Participants With Treatment Related Adverse Events | up to 8 weeks after last treatment
  Number of participants with treatment related adverse events as assessed by physical examination, vital signs, clinical laboratory values, local skin responses

SECONDARY OUTCOMES:
Percent Change from Baseline in inflammatory and non-inflammatory lesion counts | 4, 8 weeks after the last treatment
Success rate in Investigator's Global Assessment (IGA)(4wks) | 4 weeks after the last treatment
  Proportion of subjects with an assessment of clear or almost clear with at least a 2-grade improvement in IGA
Proportion of acne severity improvement as assessed with the Investigator's Global Assessment (IGA) | 4, 8 weeks after the last treatment
Change in Quality of Life of Subjects from Baseline | 4, 8 weeks after the last treatment
  Change in Quality of life will be assessed based on Acne-specific Quality of Life Questionnaire to be filled by subjects before and 4/8 weeks after last treatment

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Hospital for Skin Diseases, Chinese Academy of Medical Sciences, Nanjing, Jiangsu
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Shanghai Dermatology Hospital, Shanghai, Shanghai Municipality
  - The General Hospital of the People's Liberation Army, Beijing

IPD SHARING:
Plan to Share IPD: No